CLINICAL TRIAL: NCT06534762
Title: Efficacy and Safety of Milaberon in Combination With Standard Therapy in Advanced Solid Tumors: an Open, Multicenter, Clinical Study
Brief Title: Milaberon in Advanced Solid Tumors: an Open, Multicenter Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Minghua Ge, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Miraberon
Record Dates: First submitted 2024-07-15; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: NSCLC; SCLC; Colorectal Cancer; Pancreas Cancer; TNBC - Triple-Negative Breast Cancer; DLBCL - Diffuse Large B Cell Lymphoma; Squamous Cell Carcinoma of Head and Neck
Keywords: Lung Cancer; Pancreas Cancer; Breast Cancer; B cell lymphoma; Colorectal Cancer; Carcinoma of Head and Neck; Miraberon
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Triple Negative Breast Neoplasms; Dendritic Cell Sarcoma, Interdigitating; Squamous Cell Carcinoma of Head and Neck; Lung Neoplasms; Breast Neoplasms; Lymphoma, B-Cell | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Miraberon (Experimental): Subjects were given mirabeeron 100mg/day orally once a day in the morning until disease progression. When there are related or possible related side effects of the study drug mirabeeron, and according to NCI-CTCAE V 5.0, when subjects have more than or equal to grade 3 related toxicity, the administration should be delayed until grade 2 or lower to baseline, and the dose will be reduced by 50%, and subsequent dose increase is not allowed. If the pre-dose criteria are not met within 28 days, the drug will be permanently discontinued.
  Interventions: Biological: Mirabegron

INTERVENTIONS:
Biological: Mirabegron — To explore the efficacy and safety of milaberon combined with standard treatment in advanced solid tumors

SUMMARY:
This study is an exploratory study, and all the drugs involved are listed drugs. The dosage of mirabetron is selected according to the basis of previous research. The clinical recommend dose of this product is 50mg/day, and the dose used in this study is 100mg/day, which is larger than the clinical commonly used dose. The main adverse reactions of this product are urinary tract infection and rapid heartbeat. In the clinical study, we will focus on the urine routine and heart-related adverse events of the subjects, and deal with the adverse events in time.

Subjects were given mirabeeron 100mg/day orally once a day in the morning until disease progression. When there are related or possible related side effects of the study drug mirabeeron, and according to NCI-CTCAE V 5.0, when subjects have more than or equal to grade 3 related toxicity, the administration should be delayed until grade 2 or lower to baseline, and the dose will be reduced by 50%, and subsequent dose increase is not allowed. If the pre-dose criteria are not met within 28 days, the drug will be permanently discontinued.

DETAILED DESCRIPTION:
Cohort A non-small cell lung cancer (NSCLC):

A1 non-squamous cell carcinoma, Sintilimab or tislelizumab(3 mg/kg) pemetrexed(500mg/m2) cisplatin(75mg/m2) or carboplatin (AUC 5) q3w, 4-6 cycles of induction chemotherapy, Sintilimab or tislelizumab + pemetrexed maintenance, q3w; A2 squamous cell carcinoma, Sintilimab or tislelizumab(3 mg/kg) nab-paclitaxel (100mg/m2 d1/8/15) carboplatin (AUC 5) q3w,4-6 cycles, Sintilimab or tislelizumab maintenance, q3w; Cohort B Small cell lung cancer (SCLC) Serplulimab (4.5 mg/kg, D1) Carboplatin (AUC 5,D1) Etoposide (100 mg/m 2, D1-3),q3w, Cycle 4-6, Serplulimab maintained q3w Cohort C Colorectal cancer XELOX + bevacizumab (7.5 mg/kg,D1),q3w,8 cycles, bevacizumab + capecitabine maintenance, q3w; XELOX: oxaliplatin(130mg/m2 intravenous infusion> 2h D1), capecitabine (1000mg/m2 oral bid,D1-14),q3w; If the primary tumor is in the left colon or rectum, RAS/BRAF is wild type, cetuximab (500mg/m2,D1) + mFOLFOX6 is also admitted.

mFOLFOX6: oxaliplatin(85mg/m2, intravenous infusion 2h,D1) LV(400mg/m2, intravenous infusion 2h,D1) 5-FU (400mg, intravenous push, D1, then 1200mg/(m2 * d)X2 days continuous intravenous infusion), 12 cycles, bevacizumab + capecitabine maintenance, q3w Cohort D Pancreatic cancer GEM + nab-paclitaxel regimen, GEM(1000mg/m2) nab-paclitaxel(125mg/m2) ,D1,8, 15,q4w,6-8 cycles Adjustable GEM + nab-paclitaxel regimen, GEM(1000mg/m2) nab-paclitaxel(125mg/m2) ,D1, 8,q3w,6-8 cycles Cohort E Triple-Negative Breast Cancer TX regimen: docetaxel(75mg/m2 D1),q3w or nab-paclitaxel(100-150mg/m2 D1,qw),capecitabine(1000mg/m2 oral bid,D1-14),q3w,6-8 cycles; capecitabine maintenance, q3w (taxmen treatment sensitive) GP regimen: GEM(1000mg/m2 ,D1, 8) cisplatin(75mg/m2 ,divided into D1-3) q3w (taxane treatment failure) Cohort F Diffuse large B- cell lymphoma R-CHOP 6 cycles then R 2 cycles; R-CHOP: rituximab(375mg/m2,D0) cyclophosphamide(750mg/m2 D1),doxorubicin(40-50mg/m2,D1) vincristine(1.4mg/m2 D1 ,maximum dose 2mg) prednisone(100mg,D1-5 mg), q3w Cohort G Head and neck squamous cell carcinoma G1 Recurrent/metastatic squamous cell carcinoma of head and neck (non-nasopharyngeal carcinoma) PF: Cisplatin(100mg/m2 D1) or Carboplatin(AUC 5 D1), 5-Fu(1000mg/m2 d1-4),q3w TP: paclitaxel(175mg/m2 D1) cisplatin (75mg/m2 d1), q3w G2 Recurrent/Metastatic Nasopharyngeal Squamous Cell Carcinoma GP+Camrelizumab or Tislelizumab: cisplatin(80mg/m2 d1) gemcitabine (1000mg/m2 d1,8), then camrelizumab or tislelizumab 200mg,q3w maintenance

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in the study, sign informed consent, and have good compliance;
* 18-65 years old (including 18 and 65 years old);
* solid tumors confirmed by histology and/or cytology, and advanced metastatic tumors that are not feasible for surgical resection;
* Has not received previous systemic antitumor drug therapy for metastatic/recurrent solid tumors;
* For subjects who have previously received neoadjuvant/adjuvant therapy, it takes more than 6 months from the last treatment to relapse or progression;
* Recovery of previous treatment-related AEs to National Cancer Institute Terminology Criteria for Common Adverse Events (NCI-CTCAE)≤ Grade 1 (excluding alopecia);
* According to RECIST 1.1 standard, there is at least one measurable lesion assessed by the research center, and the measurable lesion should be a lesion that has not received local treatment such as radiotherapy (the lesion located in the region of previous radiotherapy can also be regarded as a measurable lesion that meets the requirements if progress is confirmed);
* ECOG physical condition: 0-1;
* Expected survival ≥ 12 weeks;
* The function of major organs is normal, I .e. the following criteria are met (no blood transfusion, albumin, recombinant human thrombopoietin or colony stimulating factor [CSF] treatment has been received within 14 days before the first study drug administration): blood test (absolute value of neutrophils ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin concentration ≥ 9g/dL); Liver function test (bilirubin ≤ 1.5 × ULN; aspartate aminotransferase and glutamate aminotransferase ≤ 2.5 ×ULN, AST and ALT ≤ 5 ×ULN in case of liver metastasis); renal function (serum creatinine ≤ 1.5 ×ULN, or creatinine clearance rate (CCr)≥ 60 ml/min); coagulation function, international normalized ratio (INR)≤ 1.5 ×ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT)≤ 1.5 ×ULN; thyroid function, thyroid-stimulating hormone (TSH)≤ the upper limit of normal (ULN); FT3 and FT4 levels should be examined if abnormal, and FT3 and FT4 levels are normal; (11) Women of childbearing age must have a negative serum pregnancy test within 14 days prior to treatment and be willing to use medically approved effective contraception during the study period and within 3 months after the last dose of study medication (e. g. IUDs, contraceptives or condoms; surgical sterilization is required for male subjects whose partner is a woman of childbearing age, alternatively, an effective method of contraception is recommended for the duration of the study and for 3 months after the last study dose.

Exclusion Criteria:

* Received the following treatment within 4 weeks before treatment: radiotherapy of tumor, major surgical operation or wound has not been completely healed, β3 adrenoceptor agonist and corresponding clinical research drugs;
* those who have contraindications to Miraberon: those who are allergic to Miraberon or any of its excipients;
* Active malignant tumors in the past 3 years, except for tumors participating in the study and local tumors that have been cured, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, etc;
* symptomatic brain or meningeal metastases; Severe infection (such as intravenous infusion of antibiotics, antifungals, or antivirals) within 4 weeks before treatment, or fever of unknown origin> 38.5°C during screening/first dose;
* have high blood pressure that cannot be well controlled by antihypertensive drug therapy (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
* Within 3 months before treatment, there were obvious clinical bleeding symptoms or obvious bleeding tendency (bleeding> 30 mL within 3 months, hematemesis, black stool, hematochezia), hemoptysis (fresh blood> 5 mL within 4 weeks), etc. or a venous/venous thrombotic event within 6 months prior to treatment, such as a cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; or the need for long-term anticoagulant therapy with warfarin or heparin, or the need for long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day);
* The tumor is found to invade large vascular structures during screening, such as pulmonary artery, superior vena cava or inferior vena cava, and the researchers judge that there is a greater risk of bleeding;
* Active heart disease, including myocardial infarction, severe/unstable angina pectoris, 6 months before treatment. Echocardiography left ventricular ejection fraction <50%, arrhythmia poorly controlled;
* Uncontrollable pleural effusion, pericardial effusion or ascites requiring frequent drainage after appropriate intervention;
* Presence of any active autoimmune disease or history of autoimmune disease, including but not limited to: autoimmune hepatitis, interstitial pneumonia, pulmonary fibrosis, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, thyroid function progression, decreased thyroid function; Note:(1) Subjects whose thyroid function can only be controlled by hormone replacement therapy can be included;(2) Subjects with skin diseases that do not require systemic treatment, such as vitiligo, psoriasis, alopecia, type 1 diabetes, or childhood asthma has been completely resolved, and no intervention can be included after adulthood;(3) Patients with asthma who require medical intervention with bronchodilators cannot be included;
* received treatment with live attenuated vaccine within 28 days prior to the first administration of the study drug;
* The patient has a known history of psychotropic substance abuse, alcohol abuse or drug abuse; a history of definite neurological or psychiatric disorders, including epilepsy or dementia
* tuberculosis infection history;
* known human immunodeficiency virus (HIV) infection;
* Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must exclude active HBV infection, I .e., HBV DNA positive (>1 × 104 copies/mL or> 2000 IU/mL);
* Known hepatitis C virus infection (HCV) and HCV RNA positive (>1 x 103 copies/mL), or other hepatitis, cirrhosis];
* Patients with renal injury: GFR<30 mL/min 1.73m2 or patients requiring hemodialysis
* any other medical condition, clinically significant metabolic, physical, or laboratory abnormality, which, in the investigator's judgment, would reasonably suspect that the patient has a disease or condition that is not appropriate for the study drug (e. g., having seizures requiring treatment, bladder outlet obstruction, anxiety), or would interfere with the interpretation of the study results, or place the patient in a high-risk situation, or patients considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  Overall objective tumor response rate
DLT | 3 years
  Dose-limiting toxicity

SECONDARY OUTCOMES:
DCR | 3 years
  Disease control rate
DOR | 3 years
  duration of response
TTR | 3 years
  Median time to remission
OS | 3 years
  overall survival
PFS | 3 years
  Progression free Survial

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yang, M.D., Study Director — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Zheng RS, Chen R, Han BF, Wang SM, Li L, Sun KX, Zeng HM, Wei WW, He J. [Cancer incidence and mortality in China, 2022]. Zhonghua Zhong Liu Za Zhi. 2024 Mar 23;46(3):221-231. doi: 10.3760/cma.j.cn112152-20240119-00035. Chinese. PMID 38468501
- [Background] Vasan N, Baselga J, Hyman DM. A view on drug resistance in cancer. Nature. 2019 Nov;575(7782):299-309. doi: 10.1038/s41586-019-1730-1. Epub 2019 Nov 13. PMID 31723286
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Wang R, Hu Q, Wu Y, Guan N, Han X, Guan X. Intratumoral lipid metabolic reprogramming as a pro-tumoral regulator in the tumor milieu. Biochim Biophys Acta Rev Cancer. 2023 Sep;1878(5):188962. doi: 10.1016/j.bbcan.2023.188962. Epub 2023 Aug 2. PMID 37541532
- [Background] Jin HR, Wang J, Wang ZJ, Xi MJ, Xia BH, Deng K, Yang JL. Lipid metabolic reprogramming in tumor microenvironment: from mechanisms to therapeutics. J Hematol Oncol. 2023 Sep 12;16(1):103. doi: 10.1186/s13045-023-01498-2. PMID 37700339
- [Background] Seki T, Yang Y, Sun X, Lim S, Xie S, Guo Z, Xiong W, Kuroda M, Sakaue H, Hosaka K, Jing X, Yoshihara M, Qu L, Li X, Chen Y, Cao Y. Brown-fat-mediated tumour suppression by cold-altered global metabolism. Nature. 2022 Aug;608(7922):421-428. doi: 10.1038/s41586-022-05030-3. Epub 2022 Aug 3. PMID 35922508
- [Background] O'Mara AE, Johnson JW, Linderman JD, Brychta RJ, McGehee S, Fletcher LA, Fink YA, Kapuria D, Cassimatis TM, Kelsey N, Cero C, Sater ZA, Piccinini F, Baskin AS, Leitner BP, Cai H, Millo CM, Dieckmann W, Walter M, Javitt NB, Rotman Y, Walter PJ, Ader M, Bergman RN, Herscovitch P, Chen KY, Cypess AM. Chronic mirabegron treatment increases human brown fat, HDL cholesterol, and insulin sensitivity. J Clin Invest. 2020 May 1;130(5):2209-2219. doi: 10.1172/JCI131126. PMID 31961826
- [Background] Sun X, Sui W, Mu Z, Xie S, Deng J, Li S, Seki T, Wu J, Jing X, He X, Wang Y, Li X, Yang Y, Huang P, Ge M, Cao Y. Mirabegron displays anticancer effects by globally browning adipose tissues. Nat Commun. 2023 Nov 22;14(1):7610. doi: 10.1038/s41467-023-43350-8. PMID 37993438